CLINICAL TRIAL: NCT05754125
Title: In Vivo and in Vitro Anabolic Potential of Essential Amino Acids Following Resistance Exercise
Acronym: DiEx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DiEx
Record Dates: First submitted 2023-01-31; First posted 2023-03-03 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Interventional
Keywords: Di-leucine; Branched chain amino acids; Collagen; Amino acids; anabolism; catabolism

STUDY DESIGN:
Intervention Model Description: Cross over study design; Block randomized.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither participants, investigators, or data analysts will be aware of the supplement assignment (labelled A-C) until data analysis for the primary outcome is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Di-Leucine supplement (Experimental): Participants will consume a amino acid supplement containing Di-Leucine following resistance exercise and their whole body anabolism will be determined over the subsequent 6 hours
  Interventions: Dietary Supplement: Di-Leucine Supplement
- BCAA Supplement (Experimental): Participants will consume a amino acid supplement containing branched chain amino acids (BCAA) following resistance exercise and their whole body anabolism will be determined over the subsequent hours
  Interventions: Dietary Supplement: BCAA Supplement
- Collagen Supplement (Experimental): Participants will consume a amino acid supplement containing collagen protein following resistance exercise and their whole body anabolism will be determined over the subsequent hours
  Interventions: Dietary Supplement: Collagen Supplement

INTERVENTIONS:
Dietary Supplement: Di-Leucine Supplement — Participants will consume a amino acid supplement containing Di-Leucine following resistance exercise and their whole body anabolism will be determined over the subsequent 6 hours
  Arms: Di-Leucine supplement
Dietary Supplement: BCAA Supplement — Participants will consume a amino acid supplement containing branched chain amino acids (BCAA) following resistance exercise and their whole body anabolism will be determined over the subsequent hours
  Arms: BCAA Supplement
Dietary Supplement: Collagen Supplement — Participants will consume a amino acid supplement containing Collagen protein following resistance exercise and their whole body anabolism will be determined over the subsequent hours
  Arms: Collagen Supplement

SUMMARY:
This study seeks to investigate the anabolic potential of a dileucine-enriched essential amino acid (EAA) formulation compared with a branched chain amino acid (BCAA) alternative and a collagen beverage on muscle protein anabolism and catabolism following a bout of resistance exercise training. To do this, investigators will employ a novel 'breath test' method developed in our laboratory as well as blood and urine sampling. The results of this study will allow us to better understand the anabolic potential of dileucine which could have implications for people engaging in regular resistance training (such as athletes) as well as people that need to preserve muscle mass (older people who are susceptible to anabolic resistance and sarcopenia, or muscle wasting).

ELIGIBILITY:
Inclusion Criteria:

* Trained individuals currently performing structured exercise (e.g., running, weightlifting, team-sport activity) at least 2 days per week for the previous 3 months

Exclusion Criteria:

* Inability to perform physical activity as determined by the PAR-Q
* Inability to adhere to protocol guidelines (e.g., alcohol, habitual diet)
* Regular tobacco use
* Illicit drug use (e.g., growth hormone, testosterone, etc.)
* Diagnosed medical condition under the care of a physician (e.g. type 2 diabetes)
* Inability to abstain from supplements (e.g. protein, creatine, HMB, BCAA, phosphatidic acid, etc.) at least three weeks before the trial
* Individuals on any medications known to affect protein metabolism (e.g., corticosteroids, non-steroidal anti-inflammatories, or prescription-strength acne medications)
* Participants that are amenorrheic (females only)
* On medications that may interfere with protein metabolism (e.g. anti-inflammatory drugs, hormone therapy)
* Regular tobacco use (e.g. daily use of oral or inhaled tobacco)
* Illicit drug use (e.g. growth hormone, testosterone, etc.)
* Inability to comply with the study protocol as judged by the investigators

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-21 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Whole-Body Protein Synthesis | 6 hours
  Investigators will measure the enrichment of [13CO2] in the breath by isotope ratio mass spectrometry (IRMS) in atom percent excess (APE). The measurement of carbon dioxide production (VCO2) and stable isotope tracer enrichment in the breath allows for the assessment of the rate at which amino acids are used for energy (i.e., oxidized), rather than for protein synthesis (i.e., retained in the body) by calculating the fraction of expired CO2 that contains 13C. Leucine retention (umol/kg) will then be calculated from the difference between the known amount of leucine provided (ingested) and leucine oxidation (as determined from 13CO2 breath enrichment).

SECONDARY OUTCOMES:
Urinary Measures (Muscle Protein Breakdown) | 6 hours
  Investigators will measure urinary 3-methylhistidine (3MH) as an indirect marker of muscle protein breakdown over the course of the trial (6 hours) through pooled urine collection vs baseline urine.
Murine Cell-Based Experiments (ex-vivo experiments) -hypertrophy | 60 minutes
  Investigators will use human serum obtained from fasted and fed timepoints (15, 30, 45 and 60 minutes following beverage consumption) to condition cell culture media (20% volume). To determine the effects of using fasted and/or fed 'human-conditioned' culture media on cell growth, myotube diameter (hypertrophy) will be measured via microscopy following short term (4 hours) and long-term (24 hour) incubation in the human conditioned culture media.
Murine Cell-Based Experiments (ex-vivo experiments) - Protein Synthesis | 60 minutes
  Investigators will use human serum obtained from fasted and fed timepoints (15, 30, 45 and 60 minutes following beverage consumption) to condition cell culture media (20% volume). To determine the effects of using fasted and/or fed 'human-conditioned' culture media on cell protein synthesis, puromycin incorporation (measure of protein synthesis) will be measured via western blot.
Murine Cell-Based Experiments (ex-vivo experiments) - mTORC1 Signalling | 60 minutes
  Investigators will use human serum obtained from fasted and fed timepoints (15, 30, 45 and 60 minutes following beverage consumption) to condition cell culture media (20% volume). To determine the effects of using fasted and/or fed 'human-conditioned' culture media on cell anabolic signalling mTORC1 signalling will be measured via western blot.

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Centre for High Performance Sport at the University of Toronto, Toronto, Ontario, Canada